CLINICAL TRIAL: NCT03040401
Title: A Phase I/II, Open-Label, Multicenter Study of the Safety, Efficacy and Immune Response of Histamine Dihydrochloride and Low-dose Interleukin-2 in Chronic Myelomonocytic Leukemia (CMML)
Brief Title: A Study of HDC/IL-2 Treatment in Chronic Myelomonocytic Leukemia (CMML)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); Nordic MDS Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMDSG14A
Record Dates: First submitted 2017-01-24; First posted 2017-02-02 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Leukemia, Myelomonocytic, Chronic
Keywords: CMML; Ceplene; Interleukin-2
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — Histamine; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Ceplene® and Proleukin® (Experimental): Enrolled subjects will receive histamine dihydrochloride (HDC; Ceplene®) and IL-2 (Proleukin®) subcutaneously (s.c.) twice daily (BID) in 3-week periods followed by 3 week rest periods for a total of 4 treatment cycles.
  IL-2 will be administered s.c., 1 µg/kg (=16400 IU/kg) body weight twice daily (BID) during treatment periods. Ceplene® will be administered s.c. 0.5 mg BID after IL-2 injections.
  Cohort 1 will receive only Ceplene® during the first treatment cycles and Ceplene® in combination with Proleukin® during treatment cycles 2-4.
  Interventions: Drug: Cohort 1, Ceplene® and Proleukin®
- Cohort 2: Ceplene® and Proleukin® (Experimental): Enrolled subjects will receive histamine dihydrochloride (HDC; Ceplene®) and IL-2 (Proleukin®) subcutaneously (s.c.) twice daily (BID) in 3-week periods followed by 3 week rest periods for a total of 4 treatment cycles.
  IL-2 will be administered s.c., 1 µg/kg (=16400 IU/kg) body weight twice daily (BID) during treatment periods. Ceplene® will be administered s.c. 0.5 mg BID after IL-2 injections.
  Cohort 2 will receive Ceplene® in combination with Proleukin® during all treatment cycles (1-4).
  Interventions: Drug: Cohort 2, Ceplene® and Proleukin®
- Cohort 3: Ceplene® and Proleukin® (Experimental): Enrolled subjects will receive histamine dihydrochloride (HDC; Ceplene®) and IL-2 (Proleukin®) subcutaneously (s.c.) twice daily (BID) in 3-week periods followed by 3 week rest periods for a total of 4 treatment cycles.
  IL-2 will be administered s.c., 1 µg/kg (=16400 IU/kg) body weight twice daily (BID) during treatment periods. Ceplene® will be administered s.c. 0.5 mg BID after IL-2 injections.
  Cohort 3 will receive either only Ceplene® during treatment cycles 1-4 or Ceplene® in combination with Proleukin® during treatment cycles 1-4. Treatment will be decided by the study committee based on the safety profile of treatment administered to cohort 1 and 2.
  Interventions: Drug: Cohort 3, Ceplene® and Proleukin®

INTERVENTIONS:
Drug: Cohort 1, Ceplene® and Proleukin® — Patients in Cohort 1 will be administered only Ceplene® during the first treatment cycles and Ceplene® in combination with Proleukin® during treatment cycles 2-4.
  IL-2 will be administered s.c., 1 µg/kg (=16400 IU/kg) body weight twice daily (BID) during treatment periods. Ceplene® will be administered s.c. 0.5 mg BID after IL-2.
  Arms: Cohort 1: Ceplene® and Proleukin®
Drug: Cohort 2, Ceplene® and Proleukin® — Patients in Cohort 2 will be administered Ceplene® in combination with Proleukin® during all treatment cycles 1-4.
  IL-2 will be administered s.c., 1 µg/kg (=16400 IU/kg) body weight twice daily (BID) during treatment periods. Ceplene® will be administered s.c. 0.5 mg BID after IL-2.
  Arms: Cohort 2: Ceplene® and Proleukin®
Drug: Cohort 3, Ceplene® and Proleukin® — Cohort 3 will receive either only Ceplene® during treatment cycles 1-4 or Ceplene® in combination with Proleukin® during treatment cycles 1-4. Treatment will be decided by the study committee based on the safety profile of treatment administered to cohort 1 and 2.
  IL-2 will be administered s.c., 1 µg/kg (=16400 IU/kg) body weight twice daily (BID) during treatment periods. Ceplene® will be administered s.c. 0.5 mg BID after IL-2.
  Arms: Cohort 3: Ceplene® and Proleukin®

SUMMARY:
Enrolled subjects will receive histamine dihydrochloride (HDC; Ceplene®) and/or IL-2 (Proleukin®) subcutaneously (s.c.) twice daily (BID) in 3-week periods followed by 3- or 6 week rest periods.

All subjects will be assigned to one of three consecutive cohorts, each comprising five patients.

Cohort 1 will receive HDC without IL-2 for the first treatment cycle, to enable the assessment of short-term impact of HDC alone on clonal and immunological markers. For all remaining cycles the combination of HDC and IL-2 will be given.

Cohort 2 will receive the combination of Ceplene and Proleukin in all cycles. After all patients in cohorts 1 and 2 have completed 4 treatment cycles, immunological and clinical response and toxicity will be evaluated. On the basis of the results for the first 4 cycles of cohorts 1 and 2, a third cohort of 5 patients will be enrolled receiving either the combination of HDC/IL-2 or HDC alone.

In case of a beneficial response* after 4 cycles, treatment may be continued to a total of 10 cycles. Treatment cycles 5-10 will comprise 3 weeks of treatment and 6-week rest periods.

IL-2 will be administered s.c., 1 µg/kg (=16400 IU/kg) body weight twice daily (BID) during treatment periods. Ceplene® will be administered s.c. 0.5 mg BID after IL-2. The patient or a family member/significant other will be instructed to administer injections of both study drugs to allow safe treatment at home.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of signing the informed consent form.
* CMML-1 with indication for treatment according to NMDSG guidelines*.
* Life expectancy of more than three months and ability to undergo routine outpatient evaluations for efficacy, safety, and compliance.
* The patient must be informed of the investigational nature of the study and written informed consent obtained and signed.

  * including, but not limited to increasing WBC, transfusion dependence, B-symptoms, splenomegaly.

Exclusion Criteria:

* Acute myeloid leukemia.
* CMML-2 according to WHO criteria.
* Systemic mastocytosis.
* Previous or intended allogeneic stem cell transplantation.
* Concomitant or intended cytostatic or cytoreductive therapy other than hydroxyurea (HU) *.
* ECOG performance status ≥3.
* Platelet count (TPK) <30x109/L
* NYHA class III or IV cardiac disease, hypotension or severe hypertension, vasomotor instability, serious or uncontrolled cardiac dysrhythmias (including ventricular arrhythmias) at any time, acute myocardial infarction within the past 12 months, angina pectoris or symptomatic arteriosclerotic blood vessel disease.
* Other active malignancies except in situ carcinoma of the cervix, localized squamous or basal cell carcinoma of the skin.
* Serious concurrent or recent non-malignant medical conditions which, in the opinion of the Investigator, makes the patient unsuitable for participation in this study.
* History of seizures, central nervous system disorders, stroke within the last 12 months, or psychiatric disability thought to be clinically significant in the opinion of the Investigator and adversely affecting compliance to protocol.
* Serum creatinine > 1.5 times the upper normal limit.
* Serum aminotransferase (AST), alanine transaminase (ALT) and bilirubin >2.0 times the upper normal limit
* Active autoimmune disease (including but not limited to systemic lupus, inflammatory bowel disease, and psoriasis).
* Patients with active peptic or esophageal ulcer disease or with past peptic ulcer or esophageal disease with a history or bleeding.
* Patients requiring active treatment for hypotension.
* Patients continuing systemic treatment with clonidine, steroids, and/or H2 receptor blocking agents.
* Patients with a history of histamine hypersensitivity, severe allergies to food or contrast media requiring treatment within the last five years.
* Pregnancy. Women of childbearing potential (WCBP) and males having intercourse with WCBP must agree to comply with using an effective contraceptive method for the duration of the treatment (WCBP is a sexually mature woman who is not surgically sterile or has not been naturally postmenopausal for at least 12 consecutive months).
* Nursing

  * Note that treatment with HU is allowed if treatment has been ongoing for at least 3 months prior to enrollment. The use of HU is also allowed to control myeloproliferation after starting study treatment, preferably during resting periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Adverse events as defined by CTCAE v4.03. | 3 weeks after last treatment cycle

SECONDARY OUTCOMES:
Disease progression according to IWG criteria for MDS/MPN | 3 weeks after last treatment cycle
Percentage of blasts in peripheral blood | 3 weeks after last treatment cycle
  Percentage of blasts (CD34+ cells and promonocytes) will be assessed by flow cytometry. End-of-treatment percentage will be compared to values pre-study.
Percentage of monocytes in peripheral blood | 3 weeks after last treatment cycle
  Percentage of CD14+ monocytes will be assessed by flow cytometry. End-of-treatment percentage will be compared to values pre-study.
Number of treated patients that transform to AML | 2 years after last treatment cycle
Percentage of circulating NK cells i peripheral blood | 3 weeks after last treatment cycle
  Percentage of NK cells in peripheral blood will be assessed by flow cytometry. End-of-treatment percentage will be compared to values pre-study.
Percentage of circulating CD4+ T cells i peripheral blood | 3 weeks after last treatment cycle
  Percentage of CD4+ T cells in peripheral blood will be assessed by flow cytometry. End-of-treatment percentage will be compared to values pre-study.
Percentage of circulating CD8+ T cells i peripheral blood | 3 weeks after last treatment cycle
  Percentage of CD8+ T cells in peripheral blood will be assessed by flow cytometry. End-of-treatment percentage will be compared to values pre-study.
Proportion of participants with overall survival at 2 years. | 2 years after last treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Lars Möllgård, PhD, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Huddinge, Stockholm

IPD SHARING:
Plan to Share IPD: No